CLINICAL TRIAL: NCT05663086
Title: A Randomized, Blinded, Positive-controlled Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 in Population Aged 18 Years and Above（Negative for Antibody Against COVID-19）
Brief Title: Immunogenicity and Safety of COVID-19 Vaccine in Population Aged 18 Years and Above
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: According to the development of the novel coronavirus epidemic situation and the company's R&D decision
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Collaborators: Yantai Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LYB001/CT-CHN-202
Record Dates: First submitted 2022-12-22; First posted 2022-12-23 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Population Groups; Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose vaccine (Experimental): 30μg LYB001 is to be used in the clinical trial. The number of each arm is 60.
  Interventions: Biological: One dose group; Biological: Two doses group; Biological: Aged 18-59 years; Biological: Aged 60 years old and above
- High-dose vaccine (Experimental): 60μg LYB001 is to be used in the clinical trial. The number of each arm is 60.
  Interventions: Biological: One dose group; Biological: Two doses group; Biological: Aged 18-59 years; Biological: Aged 60 years old and above
- Positive control (Active Comparator): Positive-controlled vaccine is to be used in the clinical trial. The number of each arm is 60.
  Interventions: Biological: One dose group; Biological: Two doses group; Biological: Aged 18-59 years; Biological: Aged 60 years old and above

INTERVENTIONS:
Biological: One dose group — The vaccines are to be administrated at day 0. Low dose or high dose LYB001 or positve-controlled group will be randomly assigned to receive in a 1:1:1 ratio.
Biological: Two doses group — The vaccines are to be administrated at day 0 and 28. Low dose or high dose LYB001 or positve-controlled group will be randomly assigned to receive in a 1:1:1 ratio.
Biological: Aged 18-59 years — The vaccines are to be administrated in the population of 18-59 years.Low dose or high dose LYB001 or positve-controlled group will be randomly assigned to receive in a 1:1:1 ratio.
Biological: Aged 60 years old and above — The vaccines are to be administrated in the population of 60 years old and above.Low dose or high dose LYB001 or positve-controlled group will be randomly assigned to receive in a 1:1:1 ratio.

SUMMARY:
This is a randomized, blinded, positive-controlled study to evaluate the immunogenicity and safety of Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001, in population aged 18 years old and above（negative antibody against COVID-19）. 720 subjects will be recruited in this study, including 360 in 1 dose of 30 or 60 μg group and 360 in 2 doses of 30 or 60 μg group. The age group consists of 18-59 years old and 60 years old and above.

DETAILED DESCRIPTION:
Subjects will receive 1 dose or 2 doses of LYB001, according to the immunization schedule of 0 day or 0, 28 days. The adverse events within 28 days after each vaccination will be observed. In addition, blood samples will be collected on day 0 before vaccination,and on day 7, 14, 28 and month 3, 6, 12 after full vaccination. Serum antibody levels, cellular immune responses will be analyzed to evaluate the immunogenicity and immune persistence of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 years and above who have not received COVID-19 vaccine or whose last vaccination was at least 6 months ago (at the time of screening).
* Participate the trial voluntarily and sign informed consent form.
* Subjects are willing to comply with the requirements of the clinical trial protocol and complete the study follow-up.
* Armpit temperature ≤37.0℃ on the day of enrollment.
* 2019 Novel Coronavirus (COVID-19) Antibody was negative.

Exclusion Criteria:

* Known allergy to investigational vaccine or its excipients, or previous history of anaphylactic shock or other serious adverse reactions to other vaccines
* History of severe acute respiratory syndrome (SARS) and/or Middle East respiratory syndrome (MERS) or COVID-19 infection or disease;
* Used antipyretic drugs, painkillers or anti-allergic drugs within 24 h before enrollment;
* vaccination of subunit vaccines and/or inactivated vaccines within 7 days before enrollment, or vaccination of live attenuated vaccines within 14 days before enrollment;
* Administration of blood or blood related products (including immunoglobulins) within 3 months before enrollment; or plan to use duringthe trial;
* Patients with the following diseases:

  1. Any acute disease or in the acute phase of chronic diseases within 7 days before enrollment;
  2. Congenital malformation or developmental disorder, genetic defect, severe malnutrition, etc.;
  3. History of congenital or acquired immunodeficiency or autoimmune diseases, or long-term(used continuously>14 days)use of glucocorticoid (dose ≥ 20 mg/day prednisone or equivalent dose) or other immunosuppressants within the last 6 months, yet the following situations are allowed to be included: inhaled or topical use of external steroids, or short-term use (course ≤ 14 days ) of oral corticosteroids;
  4. Positive for anti-AIDS antibody;
  5. Neurological diseases or family history (convulsion, epilepsy, encephalopathy, etc.); history of psychosis or family history;
  6. Asplenia or functional asplenia;
  7. Serious or uncontrollable cardiovascular diseases, diabetes,hematological and lymphatic diseases, immune system diseases,liver and kidney diseases, respiratory diseases, metabolism and bone diseases, or malignant tumors that need hospitalization;
  8. Contraindications of intramuscular injection and blood drawing,such as coagulation dysfunction, thrombosis or hemorrhagic diseases, or any condition that needs continuous use of anticoagulant;
  9. Severe hypertension with uncontrolled medication (at field measurement: systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg) .
* History of major surgery within 12 weeks before enrollment (judged by the investigator), or incomplete recovery after surgery, or planning major surgery during the trial;
* Participating or will participate other clinical trials during this trial;
* Any disease or condition that would pose an unacceptable risk to the subject; the subject is unable to meet the protocol requirement; will interfere with evaluation of investigational vaccine.
* Women who were breastfeeding or pregnant during the clinical study or planned to become pregnant during the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMT) of neutralizing antibody against SARS-CoV-2 wild strain | Day 14 after full vaccination.
  GMT of neutralizing antibody against SARS-CoV-2 wild strain at day 14 after full vaccination.

SECONDARY OUTCOMES:
The occurrence of adverse events | 30 mins,7 days and 28 days after each vaccination
  The occurrence of adverse events within 30 mins,7 days and 28 days after each vaccination
The occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs) | Day 0 to 12 months after dose1and dose2
  The occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs) within 12 months after dose1 and dose2
Geometric mean titers (GMT) of neutralizing antibody against SARS-CoV-2 wild strain | Day 7 , day 28 ,month 3, month 6, month 12 after full vaccination
  GMT of neutralizing antibody against SARS-CoV-2 wild strain at day 7, day 28 , month 3, month 6, month 12 after full vaccination and the difference between immunization schedule
Geometric mean fold rise(GMFR) of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs) | Day 7, day 14, day 28 , month 3, month 6, month 12 after full vaccination
  Geometric mean fold rise(GMFR) of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs) at day 7, day14, day 28 , month 3, month 6, month 12 after full vaccination and the difference between immunization schedule
Seroconversion rate of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs). | Day 7, day 14, day 28 , month 3, month 6, month 12 after full vaccination
  Seroconversion rate of neutralizing antibody against SARS-CoV-2 wild strain and variants of concern(VOCs) at day 7, day 14 ,day 28, month 3, month 6, month 12 after full vaccination and the difference between immunization schedule.
Geometric mean titers (GMT) of neutralizing antibody against variants of concern(VOCs). | Day 7, day 14, day 28 , month 3, month 6, month 12 after full vaccination
  Geometric mean titers (GMT) of neutralizing antibody against variants of concern(VOCs) at day 7, day 14 ,day 28, month 3, month 6, month 12 after full vaccination and the difference between immunization schedule.
GMT of binding antibody against S protein of SARS-CoV-2 wild strain. | Day 7, day 14, day 28 , month 3, month 6, month 12 after full vaccination
  GMT of binding antibody against S protein of SARS-CoV-2 wild strain at day 7,day 14 ,day 28,month 3, month 6, month 12 after full vaccination and the difference between immunization schedule.
Geometric mean fold rise(GMFR) of binding antibody against S protein of SARS-CoV-2 wild strain. | Day 7, day 14, day 28 , month 3, month 6, month 12 after full vaccination
  Geometric mean fold rise(GMFR) of binding antibody against S protein of SARS-CoV-2 wild strain at day 7,day 14 ,day 28,month 3, month 6, month 12 after full vaccination and the difference between immunization schedule.
Seroconversion rate of binding antibody against S protein of SARS-CoV-2 wild strain. | Day 7, day 14, day 28 , month 3, month 6, month 12 after full vaccination
  Seroconversion rate of binding antibody against S protein of SARS-CoV-2 wild strain at day 7,day 14 ,day 28,month 3, month 6, month 12 after full vaccination and the difference between immunization schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China